CLINICAL TRIAL: NCT01782820
Title: Influence of a Single Dose Dexamethasone on the Time Course of Neuromuscular Blockade of Rocuronium
Status: Completed | Type: Observational
Sponsor: Kreiskrankenhaus Dormagen (Other)
Responsible Party: Sponsor
Other Study IDs: dexarelax
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Neuromuscular Block, Dexamethasone; Neuromuscular Block, Recovery

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- dexamethasone late: dexamethasone during induction of anesthesia
- no dexamethasone: no dexamethasone during measurements
- dexamethasone early: dexamethasone before induction of anesthesia

SUMMARY:
The aim of the present study is to compare the time course of a neuromuscular block in patients receiving dexamethasone 8 mg in order to reduce postoperative nausea or vomiting several hours before surgery with patients receiving the drug immediately before induction of anaesthesia and patients without a dexamethasone prophylaxis. The primary end point is the time from start of injection of rocuronium until recovery to a train of four ratio (TOF ratio) of 0.9.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 65 years,
* American Society of Anesthesiologists Physical Status I or II,
* 50-90 kg body weight,
* undergoing elective laparoscopic gynaecological surgery in general anaesthesia necessitating intraoperative neuromuscular blockade.

Exclusion Criteria:

* expected difficulties with endotracheal intubation (history of difficult intubation,
* reduced opening of the mouth (< 2cm), and Mallampati Score of 4),
* increased risk of pulmonary aspiration (gastrooesophageal reflux, full stomach, intestinal obstruction),
* known allergies to the drugs tested,
* pregnancy,
* neuromuscular disorders,
* intake of drugs affecting neuromuscular blockade, such as furosemide, magnesium or cephalosporins,
* hepatic-or renal insufficiency.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of a primary care clinic undergoing elective gynecologic abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
the time from start of injection of rocuronium until recovery to a train of four ratio (TOF ratio) of 0.9. | one hour

CONTACTS AND LOCATIONS:
Locations (1):
- Kreiskrankenhaus Dormagen, Dormagen, Germany

REFERENCES:
- [Derived] Soltesz S, Fraisl P, Noe KG, Hinkelbein J, Mellinghoff H, Mencke T. Dexamethasone decreases the duration of rocuronium-induced neuromuscular block: a randomised controlled study. Eur J Anaesthesiol. 2014 Aug;31(8):417-22. doi: 10.1097/EJA.0b013e328365c9ee. PMID 24136379